CLINICAL TRIAL: NCT07306247
Title: Multicenter Prospective Non-randomized Controlled Study of Ella Photodynamic Therapy for Cervical Low-grade Squamous Intraepithelial Lesions With HPV16/18 Infection
Brief Title: Multicenter Prospective Non-randomized Controlled Study of ALA-PDT for LSIL With HPV16/18 Infection
Acronym: PDT for LSIL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Women's Hospital School Of Medicine Zhejiang University (Other); First People's Hospital of Hangzhou (Other); First Affiliated Hospital of Ningbo University (Network); Shaoxing People's Hospital (Other); Linping First People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1380
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: HPV-16/18; Photodynamic Therapy (PDT); LSIL, Low Grade Squamous Intraepithelial Lesion
Keywords: cervical low-grade squamous intraepithelial lesions; aminolevulinic acid-mediated photodynamic therapy; efficacy; human papillomavirus
MeSH Terms: conditions — Squamous Intraepithelial Lesions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALA-PDT Group (Experimental): ALA-PDT administered every 7-14 days for a total of 3-6 sessions.
  Interventions: Procedure: ALA-PDT
- Observation Group (No Intervention): Observation and follow-up

INTERVENTIONS:
Procedure: ALA-PDT — Photosensitizer is applied to the cervical canal and cervix, followed by light irradiation, repeated every 7-14 days for 3-6 sessions.
  Arms: ALA-PDT Group

SUMMARY:
This multicenter, prospective trial assesses ALA-PDT versus observation for efficacy and safety in treating cervical LSIL with HPV16/18 infection.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, concurrent, non-randomized controlled clinical trial designed to evaluate the clinical efficacy of ALA-PDT treatment compared with observation and follow-up in patients with cervical low-grade squamous intraepithelial lesion (LSIL) associated with HPV16/18 infection. The primary outcome is the cervical lesion reversal rate. Secondary outcomes include HPV16/18 clearance rate and time to clearance, as well as improvements in cervical ectropion and vaginal microenvironment. Additionally, lesion progression rate and recurrence rate will be monitored in both groups. Safety, tolerability, patient-reported quality of life, and treatment satisfaction are also assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 20-60 years, understands study procedures and consents to participate;
2. HPV 16 or 18 positive;
3. Colposcopy-guided cervical biopsy within 3 months showing LSIL;
4. Provides written informed consent.

Exclusion Criteria:

1. Cytology showing ASC-H, HSIL, AGC, or AIS; or evidence of malignant cells on cytology/histology, or suspicion of malignancy or invasive cancer;
2. Colposcopy findings suggestive of invasive cancer or lesion extension to the vaginal wall;
3. Severe pelvic, cervical, or other gynecological inflammatory conditions identified clinically;
4. Undiagnosed vaginal bleeding;
5. Active allergic disease, porphyria, or history of allergy to the study drug or structurally similar agents;
6. Severe cardiovascular, neurological, psychiatric, endocrine, hepatic, or hematologic disorders; known immunodeficiency; long-term glucocorticoid or immunosuppressant use; active autoimmune disease; or other malignancies;
7. Pregnant or breastfeeding women;
8. History of hysterectomy, cervical cancer treatment, or cervical excision/ablation within 6 months (e.g., conization, LEEP, laser);
9. Use of interferon or antiviral therapy within 3 months;
10. Any other condition deemed unsuitable for participation by the investigator.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cervical lesion regression rate | 6 months
  Proportion of patients with normal histopathology on colposcopy-guided biopsy or NILM cytology, plus negative HPV test, at 6 months post-treatment.

SECONDARY OUTCOMES:
HPV clearance rate | 2 years
  HPV clearance rates at 3, 6, 9, 12, and 24 months post-treatment
Cervical lesion regression rate | 2 years
  Proportion of patients with normal colposcopy-guided cervical biopsy histopathology, or NILM cytology plus negative HPV test, at 12 and 24 months.

OTHER OUTCOMES:
Adverse events | 2 years
  Record post-treatment bleeding, pain, and photosensitivity.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang
  - First People's Hospital of Hangzhou, Hangzhou, Zhejiang
  - Hangzhou Linping District first People's Hospital, Hangzhou, Zhejiang
  - First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kajdanski E. Receptarum sinensium liber of Michael Boym. Janus. 1986-1990;73:105-19. No abstract available. PMID 11622471
- [Result] Wang X, You L, Zhang W, Ma Y, Tang Y, Xu W. Evaluation of 5-aminolevulinic acid-mediated photodynamic therapy on cervical low-grade squamous intraepithelial lesions with high-risk HPV infection. Photodiagnosis Photodyn Ther. 2022 Jun;38:102807. doi: 10.1016/j.pdpdt.2022.102807. Epub 2022 Mar 11. PMID 35288319
- [Result] Qiu L, Li J, Chen F, Wang Y, Wang Y, Wang X, Lv Q, Li C, Li M, Yang Q, Wu D, Zhang Y, Zhang Y, Zhang M, Zhang Y, Qie M, Zhou H, Zhou J, Zhao W, Xia B, Liang X, Cai Y, Teng Y, Huang Z, Sui L, Wei L, Di W. Chinese expert consensus on the clinical applications of aminolevulinic acid-based photodynamic therapy in female lower genital tract diseases (2022). Photodiagnosis Photodyn Ther. 2022 Sep;39:102993. doi: 10.1016/j.pdpdt.2022.102993. Epub 2022 Jul 1. PMID 35781093
- [Result] Wang X, Xu X, Ma Y, Tang Y, Huang Z. Comparative Study of 5-Aminolevulinic Acid-Mediated Photodynamic Therapy and the Loop Electrosurgical Excision Procedure for the Treatment of Cervical High-Grade Squamous Intraepithelial Lesions. Pharmaceutics. 2024 May 20;16(5):686. doi: 10.3390/pharmaceutics16050686. PMID 38794347
- [Result] Persson M, Elfstrom KM, Olsson SE, Dillner J, Andersson S. Minor Cytological Abnormalities and up to 7-Year Risk for Subsequent High-Grade Lesions by HPV Type. PLoS One. 2015 Jun 17;10(6):e0127444. doi: 10.1371/journal.pone.0127444. eCollection 2015. PMID 26083247
- [Result] Kusakabe M, Taguchi A, Sone K, Mori M, Osuga Y. Carcinogenesis and management of human papillomavirus-associated cervical cancer. Int J Clin Oncol. 2023 Aug;28(8):965-974. doi: 10.1007/s10147-023-02337-7. Epub 2023 Jun 9. PMID 37294390
- [Result] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751